CLINICAL TRIAL: NCT05129943
Title: Efficacy of Active and Passive Virtual Reality Distraction During Local Anesthesia in Children
Brief Title: Efficacy of VR Distraction During Local Anesthesia in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tishreen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VR distraction in children
Record Dates: First submitted 2021-11-11; First posted 2021-11-22 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-02

CONDITIONS: Virtual Reality; Anesthesia, Local; Pain
Keywords: virtual reality; local anesthesia; pain; distraction
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: the participants will be divided into ( active distraction group) and ( passive distraction group )
Who Masked: Investigator, Outcomes Assessor
Masking Description: the participants will carry the controller with a box to hide the controller (to keep the outcomes assessor blinded) and wear the VR device by an assistant ( to keep investigator blinded).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active distraction group (Active Comparator): local anesthesia with video game using VR device
  Interventions: Device: active distraction
- passive distraction group (Active Comparator): local anesthesia with cartoon video using VR device
  Interventions: Device: passive distraction

INTERVENTIONS:
Device: active distraction — The subject receives the injection of local anesthesia while playing a game on a mobile phone mounted on the VR device using a PS4 controller.
  Arms: active distraction group
Device: passive distraction — The subject receives the injection of local anesthesia while watching a cartoon on a mobile phone mounted on the VR device.
  Arms: passive distraction group

SUMMARY:
The aim of this study is to compare between active distraction (video game) and passive distraction (cartoon video) using a Virtual Reality ( VR ) device, in reducing injection pain and anxiety associated with local anesthesia in children.

DETAILED DESCRIPTION:
This comparative study is a double blinded controlled randomized clinical trial which includes 82 healthy 6-10 years old children with positive and definitely positive behavior according to Frankl Rating Scale with no known allergy to local anesthesia, no emergency dental treatment, no previous treatment from the same researcher and no previous experience in using the Virtual Reality ( VR ) device.

the participants will be allocated and treated at department of pediatric dentistry, faculty of dentistry, Tishreen university and a written consent will be obtained from the parents.

The random-numbers table will be used to divide 82 participants in to two groups:

1. The active distraction group, which will be receiving the injection of local anesthesia while using the VR device with a video game and a Play Station 4 ( PS4 ) controller.
2. The passive distraction group, which will be receiving the injection of local anesthesia while using VR device watching a cartoon video.

All the participants will receive an inferior alveolar nerve block with semi supine position.

ELIGIBILITY:
Inclusion Criteria:

* healthy children need a simple treatment for temporary teeth in the mandibular jaw
* children with positive and definitely positive behavior according to frankl behavior classification
* children with no known allergy to local anesthesia
* children with no previous treatment from the same researcher
* children with no previous experience in using the VR device

Exclusion Criteria:

* children with negative and definitely negative behavior according to frankl behavior classification
* children with known allergy to local anesthesia
* children with emergency dental treatment in the mandibular jaw
* children with previous treatment from the same researcher

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
dental pain | during the injection of local anesthesia
  evaluated by outcome assessor using the Faces, Legs, Activity, Cry, Consolability Behavioral Pain Rating Scale ( FLACC scale ) ( a behavioral pain assessment scale which has five criteria face, legs, activity, cry, consolability ,which are each assigned a score of 0, 1 or 2.Total score of scale is summed in range 0 to 10, where: 0=relaxed and comfortable; 1-3=mild discomfort; 4-6=moderate pain; 7-10=severe pain).
dental pain | Immediately after the injection of local anesthesia
  self assessment pain by the children using Wong-Baker faces pain rating scale (a scale shows a series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10,which represents "hurts like the worst pain imaginable" )

SECONDARY OUTCOMES:
dental pain and anxiety | during the injection of local anesthesia
  using mi band 3 to recording the pulse

CONTACTS AND LOCATIONS:
Overall Officials: oula kara Mohammed, DDS, Principal Investigator — Tishreen University; Nabih Raslan, Dr., Study Chair — Tishreen University
Locations (1):
- Tishreen university, Latakia, Syria